CLINICAL TRIAL: NCT03866707
Title: Epigenetic and Metabolomic Changes in Childhood Cancer Survivors as a Late Effect of Treatment - a Pilot Study
Brief Title: Epigenetic and Metabolomic Changes in Childhood Cancer Survivors
Status: Terminated | Type: Observational
Why Stopped: PI left institution, study will not resume and considered complete
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00048882; CCCWFU 01118 (Other: Wake Forest University Health Science)
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Childhood Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: One-time blood draw — Subjects will have a one-time blood draw of 5-10mL. Quantity of blood drawn for study and routine care will not exceed the maximum safe blood volume for subject size.
  Evaluation of CpG methylation sites will be completed using the MethylationEPIC BeadChip (Infinium) microarray. This covers over 850,000 CpG methylation sites and is available in the investigator's Genomics Core Facility. Dr. Langefeld has analyzed numerous methylation studies, both array-based and next generation sequencing.
  Metabolomic analysis will be performed by mass spectrometry when funds are available.
Other: Evaluation of CpG methylation — Evaluation of CpG methylation sites will be completed using the MethylationEPIC BeadChip (Infinium) microarray.
Other: Metabolomic analysis — Metabolomic analysis will be performed by mass spectrometry when funds are available.

SUMMARY:
The purpose of this research study is to try and identify markers in childhood cancer survivors to help predict if they will develop late effects from their cancer treatment.

DETAILED DESCRIPTION:
This is a pilot study to obtain preliminary data that will be used to apply for a larger grant to fund the full study with an adequate sample size for analysis.

Specific Aim 1. What are the epigenetic differences between children treated for childhood cancers and healthy controls matched for age, sex, ethnicity, geographic region, and tanner stage.

Specific Aim 2. Compare the metabolomic differences between children treated for childhood cancers and healthy controls matched for age, sex, ethnicity, geographic region, and tanner stage.

ELIGIBILITY:
Inclusion Criteria:

* Childhood cancer survivors age 1-18 years old who received intensive treatment which included anthracycline and/or alkylating agent chemotherapy.
* Diseases which will be eligible include, high risk or very high risk acute lymphoblastic leukemia, acute myeloid leukemia, Hodgkin lymphoma, non-Hodgkin lymphoma, sarcomas.

Healthy controls:

• Healthy controls are defined as children ages 1-18 years old who are free from diseases or medical conditions that might be affected by or have an impact on this research study. Healthy controls will be matched with patients for age, sex, ethnicity, geographic region, and tanner stage, since it is known that these factors can affect the epigenetic signature of an individual. Controls will already be having blood drawn as part of their routine care.

Exclusion Criteria:

Cancer survivors:

• Patients who have received a bone marrow transplant will not be eligible.

Healthy controls:

• Age, sex, ethnicity, geographic region, and tanner stage matched controls with any acute or chronic disease will be excluded.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators propose to evaluate 8 patients who have been treated for childhood cancer and are at least 6 months off therapy. Because methylation patterns are known to change in different populations, 8 control patients matched for age, sex, and tanner stage will also be evaluated. Because of their under representation in clinical research, initially the investigators will recruit cancer survivors and controls of Caucasian Hispanic ethnicity from the same geographic region (i.e., Piedmont region of North Carolina).
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Epigenetic Testing | Over 9 months
  Baseline and follow-up differences (predictor) in CpG methylation at sites on the EPIC array will be compared between subjects and controls (outcomes). Samples will be evaluated using the Infinium Methylation EPIC BeadChip microarray. This evaluates over 850,000 CpG methylation sites. The proportion of methylation for each site is based on the ratio of the fluorescence intensity of the methylated versus the combined methylated and unmethylated probes (referred to as the β value), and will be determined with GenomeStudio (Illumina, Inc.). For analysis, all β values will be converted to M values, where M is the log2 ratio of the methylated probe intensity to the unmethylated probe intensity.
Metabolomic testing | Over 9 months
  Metabolic profiling will be done on serum using ultrahigh-performance liquid-phase chromatography and gas-chromatography separation, coupled with tandem mass spectrometry (UHPLC/MS/MS2 and GC/MS, respectively) at Metabolon, Inc. (Durham, NC, USA) using established procedures and technology. (10) samples will be collected at three time points based on disease type and will be flash frozen in liquid nitrogen after collection and stored at -80°C to ensure sample stability.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Buckley, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States